CLINICAL TRIAL: NCT02481414
Title: A Phase II Clinical Trial of PepCan Randomized and Double-Blinded to Two Therapy Arms for Treating Cervical High-Grade Squamous Intraepithelial Lesions
Brief Title: A Clinical Trial of PepCan to Two Therapy Arms for Treating Cervical High-Grade Squamous Intraepithelial Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202790
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: HSIL, CIN II/III
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions

STUDY DESIGN:
Intervention Model Description: PepCan or Candin randomized at a 1:1 ratio in a double-blinded design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PepCan (Experimental): Four injections (one every 3 weeks) of PepCan
  Interventions: Biological: PepCan
- Candin (Active Comparator): Four injections (one every 3 weeks) of Candin
  Interventions: Biological: Candin®

INTERVENTIONS:
Biological: PepCan — 50 μg peptide + 0.3 mL Candin® per dose administered intradermally in the extremities
  Other Names: HPV 16 E6 peptides combined with Candin®
  Arms: PepCan
Biological: Candin® — 0.3 mL Candin® per dose administered intradermally in the extremities
  Other Names: Candida skin testing reagent
  Arms: Candin

SUMMARY:
This is a Phase II study to evaluate the efficacy and safety of a human papilloma virus (HPV) therapeutic vaccine called PepCan (HPV 16 E6 peptides combined with Candida skin testing reagent called Candin®) in adult females over a 12 month time period. As the results from the Phase I trial demonstrated some efficacy against non-16 HPV types, Candin alone will also be tested. Therefore, there will be two treatment arms: (1) PepCan and (2) Candin. Subjects found to be eligible for vaccination will be randomized in a double-blinded fashion at a 1:1 ratio. Each participant will be receiving injections four times with three weeks between injections. Clinical and virological responses will be assessed at 6 and 12 months. Safety will be assessed from the time of enrollment to 12 Month Visit. Immunological assessments will be made at 4 time points (prevaccination, after 2 injections, 6 month after 4 injections and 12 months after 4 vaccinations).

DETAILED DESCRIPTION:
This is a single site Phase II clinical trial of PepCan for treating women with biopsy-proven HSILs (High Grade Intraepithelial Lesions) randomized and double-blinded to two treatment arms. Half of the subjects will receive PepCan, and the other half will receive Candin® alone. The study design closely resembles the latest guidelines for treating young women with HSIL. Study subjects will be patients attending the University of Arkansas for Medical Sciences (UAMS) Obstetrics and Gynecology Clinics with untreated biopsy-proven HSILs and patients referred from other clinics. Four injections (one every 3 weeks) of PepCan or Candin® will be intradermally administered in the extremities. Clinical response will be assessed by comparison of colposcopy-guided biopsy results obtained prior to vaccination and at 12-Month Visit. Safety will be monitored from the time of enrollment through the 12-Month Visit. Blood will be drawn for laboratory testing and immunological analyses ("blood test") prior to injection, after the second vaccination, 6 months after the fourth vaccination, and 12 months after the fourth vaccination. Blood will be drawn to aid T-cell analyses ("blood draw") after the first and third vaccinations, and possibly at the Optional Follow-Up and/or Optional Loop Electrosurgical Excision Procedure (LEEP) visits. HPV-DNA testing will be performed at Screening and 6- and 12-Month Visits. If a subject has persistent HSIL at the 12-Month Visit or if a subject is withdrawn due to excessive toxicity, she will be given an option to return for a LEEP visit. Alternatively, she may choose to exit the study and be followed by a gynecologist for up to 2 years of observation as recommended before surgical treatment

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years
* Had recent (≤ 60 days) Pap smear result consistent with high grade squamous intraepithelial lesion (HSIL) or "cannot rule out HSIL" or HSIL on colposcopy-guided biopsy
* Untreated for HSIL or "Cannot rule out HSIL"
* Able to provide informed consent
* Willingness and able to comply with the requirements of the protocol

Exclusion Criteria:

* History of disease or treatment causing immunosuppression (e.g., cancer, human immunodeficiency virus (HIV), organ transplant, autoimmune disease)
* Being pregnant or attempting to be pregnant within the period of study participation
* Breast feeding or planning to breast feed within the period of study participation
* Allergy to Candida antigen
* History of severe asthma requiring emergency room visit or hospitalization within the past 5 years
* History of invasive squamous cell carcinoma of the cervix
* History of having received PepCan
* If in the opinion of the Principal Investigator or other Investigators, it is not in the best interest of the patient to enter this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayumi N Nakagawa, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PepCan | Candin
Started | 39 | 42
Completed | 35 | 41
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PepCan | Candin | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Customized [Mean (Standard Deviation); unit: years] | 31.3 (6.4) | 31.4 (6.1) | 31.3 (6.2)
Age, Customized [Mean (Full Range); unit: years] | 31.3 [21.5 to 45.1] | 31.4 [22.4 to 43.6] | 31.3 [21.5 to 45.1]
Age, Customized [Count of Participants; unit: Participants] — Number of Participants with Age <25 years and ≥25 years
  Participants
    <25 years - number (no.) | 6 | 9 | 15
    ≥25 years - number (no.) | 33 | 33 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Number of participants who are Hispanic of Latino, Not Hispanic or Latino, or Unknown or Not Reported
  Participants
    Hispanic or Latino | 11 | 12 | 23
    Not Hispanic or Latino | 28 | 30 | 58
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of participants who are race Caucasian, African American, or Other
  Participants
    Caucasian | 34 | 37 | 71
    African American | 4 | 4 | 8
    Other | 1 | 1 | 2
Histological Diagnosis at Study Entry [Count of Participants; unit: Participants] — Histological grade determined using cervical biopsies at study entry.
  CIN2 is moderate dysplasia and CIN3 is serve dysplasia. CIN2/3 is in between moderate and server dysplasia.
  Participants
    CIN3 and CIN2/3 | 29 | 26 | 55
    CIN2 | 10 | 16 | 26
Number (No.) of cervical quadrants [Mean (Standard Deviation); unit: cervical quadrants] — Mean Number (No.) of cervical quadrants
  cervical quadrants | 1.89 (1.06) | 2.05 (1.02) | 1.97 (1.04)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Mean body mass index in kg/m^2 for participants
  kg/m^2 | 27.3 (6.2) | 29.1 (7.3) | 28.3 (6.8)
Albumin < 3.5 g/dL [Count of Participants; unit: Participants] — Number of Participants with Albumin < 3.5 g/dL
  Participants | 1 | 3 | 4
Total protein < 6.4 g/dL [Count of Participants; unit: Participants] — Number of Participants with Total protein < 6.4 g/dL
  Participants | 3 | 5 | 8
Human papillomavirus (HPV) prophylactic vaccine [Count of Participants; unit: Participants] — Number of Participants with Human papillomavirus (HPV) prophylactic vaccine
  Participants | 7 | 7 | 14
Any college [Count of Participants; unit: Participants] — Number of Participants with Any college
  Participants | 20 | 20 | 40
Any children [Count of Participants; unit: Participants] — Number of Participants with Any children
  Participants | 27 | 27 | 54
≥ 5 sexual partners [Count of Participants; unit: Participants] — Number of Participants with ≥ 5 sexual partners
  Participants | 19 | 30 | 49
Ever smoked [Count of Participants; unit: Participants] — Number of Participants who has Ever smoked
  Participants | 18 | 15 | 33
Currently smoke [Count of Participants; unit: Participants] — Number of Participants who Currently smoke
  Participants | 8 | 9 | 17
Ever used oral contraceptives [Count of Participants; unit: Participants] | 27 | 32 | 59
Currently use oral contraceptives [Count of Participants; unit: Participants] — Number of participants who Currently use oral contraceptives
  Participants | 6 | 15 | 21
Number (No.) of cervical quadrants [Count of Participants; unit: Participants] — Number of participants with cervical quadrants > 2 Quadrants and ≤ 2 Quadrants. The cervical quadrant data weas not available from two of the participants (one in PepCan group and other in Candin Group).
  Participants
    >2 quadrants | 9 | 11 | 20
    ≤2 quadrants | 29 | 30 | 59
    Data not available | 1 | 1 | 2
Body mass index [Count of Participants; unit: Participants] — Number of participants who how have body mass index of ≥25 kg/m^2 - <30 kg/m^2 and ≥30 kg/m^2
  Participants
    ≥25 kg/m^2 - <30 kg/m^2 | 10 | 7 | 17
    ≥30 kg/m^2 | 11 | 19 | 30
    <25 kg/m^2 | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complete Response With the Intention-to-treat (ITT) Analysis
Description: Histological regression of moderate/severe cervical dysplasia to absence of cervical dysplasia assessed using biopsies (stringent)
Time Frame: 15 months from time of last vaccination
Population: ITT (subjects who were eligible and randomized)
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan | Candin
Number analyzed (Participants) | 39 | 42
Participants | 12 | 20

2. Primary Outcome: Number of Subjects With Complete Response With the Per-protocol Analysis
Description: Histological regression of moderate/severe cervical dysplasia to absence of cervical dysplasia assessed using biopsies (stringent)".
Time Frame: 15 months from time of last vaccination
Population: Per-protocol (subjects who completed the 12-month visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan | Candin
Number analyzed (Participants) | 24 | 29
Participants | 11 | 18

3. Primary Outcome: Number of Subjects With Complete and Partial Responses With the ITT Analysis
Description: Histological regression of moderate/severe cervical dysplasia to mild dysplasia/no dysplasia (lenient) assessed using biopsies, likely avoiding a need for surgery
Time Frame: 15 months from time of last vaccination
Population: ITT (subjects who were eligible and randomized)
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan | Candin
Number analyzed (Participants) | 39 | 42
Participants | 15 | 24

4. Primary Outcome: Number of Subjects With Complete and Partial Responses With the Per-protocol Analysis
Description: as for outcome 3
Time Frame: 15 months from time of last vaccination
Population: Per-protocol (subjects who completed the 12-month visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PepCan | Candin
Number analyzed (Participants) | 24 | 29
Participants | 13 | 22

5. Secondary Outcome: Safety Assessed by Injection-related Adverse Events (AEs)
Description: Injection-related AEs occurring in >5% of injections
Time Frame: 15 months from time of last vaccination
Population: Number of Injections for ITT (subjects who were eligible and randomized)
Measure: Number; unit: Adverse Events
Units Other Than Participants: Number of Injections
Arm/Group | PepCan | Candin
Number analyzed (Participants) | 39 | 42
Number analyzed (Number of Injections) | 152 | 164
Adverse Events
  Fever : Grade 1 | 9 | 3
  Fever : Grade 2 | 1 | 0
  Fever : All Grades | 10 | 3
  Headache : Grade 1 | 13 | 15
  Headache : Grade 2 | 4 | 3
  Headache : All Grades | 17 | 18
  Injection site reaction, < 24 h : Grade 1 | 63 | 58
  Injection site reaction, < 24 h : Grade 2 | 25 | 31
  Injection site reaction, < 24 h : All Grades | 88 | 89
  Myalgia : Grade 1 | 35 | 9
  Myalgia : Grade 2 | 2 | 1
  Myalgia : All Grades | 37 | 10
  Nausea : Grade 1 | 19 | 18
  Nausea : Grade 2 | 0 | 0
  Nausea : All Grades | 19 | 18
  Injection site reaction, ≥ 24 h : Grade 1 | 23 | 39
  Injection site reaction, ≥ 24 h : Grade 2 | 31 | 18
  Injection site reaction, ≥ 24 h : All Grades | 54 | 57

ADVERSE EVENTS:
Time Frame: Time of enrollment until 15 months from time of last vaccination, approximately 18 months
Arm/Group | PepCan | Candin
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/39 | 2/42
Other Adverse Events (participants affected / at risk) | 37/39 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PepCan (N=39) | Candin (N=42)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Fetal Death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Psychiatric Disorders - Other Specify (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PepCan (N=39) | Candin (N=42)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 7 (8)
Chest Pain - Cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (3)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Eye Disorders 0 Other, Specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (6) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (31) | 12 (22)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Vomitting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 3 (4) | 4 (4)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (9) | 7 (9)
Fever (General disorders) | 10 (14) | 4 (5)
Flu-like Symptoms (General disorders) | 6 (8) | 4 (5)
Injection Site Reaction (General disorders) | 34 (142) | 38 (146)
Localized Edema (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (2)
Pain (General disorders) | 3 (8) | 4 (4)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 6 (9) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 5 (7) | 4 (4)
Vaginal Infection (Infections and infestations) | 4 (5) | 5 (5)
Infections and Infestations - Others, Specify (Infections and infestations) | 3 (3) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 8 (8) | 5 (5)
Alkaline Phosphatase Increased (Investigations) | 2 (2) | 1 (1)
Blood Bilirubin Increased (Investigations) | 2 (2) | 1 (1)
Creatinine Increased (Investigations) | 5 (5) | 3 (4)
Hemoglobin Increased (Investigations) | 3 (4) | 2 (2)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (2)
Weight Loss (Investigations) | 1 (1) | 0 (0)
White Blood Cell Decreased (Investigations) | 1 (2) | 2 (2)
Investigations - Other, Specify (Investigations) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 9 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7) | 10 (12)
Hyponatremia (Metabolism and nutrition disorders) | 5 (7) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (44) | 9 (12)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and Connective Tissue Disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Concentration Impairement (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (8) | 5 (10)
Headache (Nervous system disorders) | 10 (25) | 12 (25)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Nervous System Disorders - Other, Specify (Nervous system disorders) | 1 (1) | 0 (0)
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (6) | 3 (3)
Depression (Psychiatric disorders) | 2 (3) | 2 (3)
Psychiatric Disorders - Other, Specify (Psychiatric disorders) | 3 (4) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal and Urinary Disorders - Other, Specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Irregular Menstruation (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal Inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginismus (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive System and Breast Disorders - Other, Specify (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Hot Flashes (Vascular disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 6 (7) | 7 (7)
Skin Infection (Infections and infestations) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT02481414/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02481414/SAP_002.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT02481414/ICF_000.pdf